CLINICAL TRIAL: NCT02526563
Title: Serum Ropivacaine Concentrations in Pediatric Patients Receiving Continuous Wound Catheter Analgesia
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Franklyn Cladis, MD, University of Pittsburgh
Other Study IDs: PRO14110169
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Alveolar Bone Grafting; Alveolar Cleft Grafting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Iliac crest wound catheter group: These patients will receive an iliac crest wound catheter after an iliac crest bone harvest to repair a palatal defect. This catheter is part of standard of care. This study will collect blood to measure unbound ropivicaine levels.
  Interventions: Procedure: ropivicaine

INTERVENTIONS:
Procedure: ropivicaine — Blood draws to measure serum ropivicaine

SUMMARY:
The primary investigators in this study plan to investigate serum concentrations of ropivacaine in pediatric patients who already receive as standard of care a continuous wound catheter after an iliac crest alveolar bone graft harvest for completion of a previous cleft palate repair.

The goals of this study are 1) to determine serum concentrations (free, unbound) of ropivacaine 2) To evaluate pain scores during the perioperative period to determine efficacy of wound catheters for postoperative analgesia for iliac crest bone graft harvest.

DETAILED DESCRIPTION:
There have been numerous investigations of serum concentration of ropivicaine using wound catheters in adults. These studies have revealed that wound catheters provide effective analgesia without toxic levels of serum ropivicaine. Our current proposal is different for two reasons. One, the investigators will be investigating the serum levels of ropivacaine in pediatric patients. There are currently no studies investigating the efficacy of this technique in the pediatric population. Two, the wound catheter currently being placed by Dr Losee (and plastic surgeons in other pediatric centers) as part of standard of care is different from other wound catheters. Most wound catheters described in the literature are placed in the surgical wound between muscle and facial planes. The catheter placed by Dr Losee for his routine postoperative pain control is placed adjacent to the periosteum and adjacent to the bone harvest site. Dr Losee has been performing this technique as part of standard patient care and it appears to provide excellent analgesia without side effects from the ropivacaine. However, it is unknown what effect this location has on serum plasma levels of ropivacaine. Measuring unbound ropivacaine will help define whether or not these wound catheters maintain the serum ropivacaine levels below, near, or above toxic levels. Pediatric studies have investigated the serum ropivacaine levels during epidural infusions and peripheral nerve blocks. This local anesthetic is safe as long as the administration is limited to weight based limits. For continuous infusions, ropivacaine should not be administered at a greater rate than 0.4 -0.5 mg/kg/hr. The wound catheters for The Childrens Hospital of Pittsburgh Plastic Surgery service are administered at 0.25 mg/kg/hr. Ropivacaine is the local anesthetic of choice for many pediatric hospitals and for the Acute Interventional Pediatric Pain Service at the Children's Hospital of Pittsburgh because it appears to have a slight safety advantage over bupivacaine. Ropivacaine does not bind sodium channels as avidly as bupivacaine and therefore may not be as cadiac toxic. However, the location of the catheter can alter absorption and may alter plasma levels. Currently there is no data for pediatric iliac crest wound catheters. Since this technique is already a standard of care here at this center, we plan to measure serum ropivacaine levels to define these values.

It is important to understand the dosages currently being used in this pediatric population and the effects on serum local anesthetic levels. When local anesthetic is infused through an epidural, peripheral nerve block, or wound catheter, there is an elevation in local anesthetic plasma levels in the patient. The plasma levels depend on the dose, concentration and location of the catheter. Current literature has defined the plasma levels obtained during continuous infusions of local anesthetic through wound catheters in adults. Safe infusion rates have been defined for adult catheters. This data does not exist for wound catheters in pediatric patients and this study will begin to define these limits. In particular, the catheter currently being placed as standard of care at The Children's Hospital of Pittsburgh is periostial and it is unknown what effect this location has on serum ropivacaine levels

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria is any patient age ranging from 5 to 18 years of age that is scheduled for an iliac crest bone harvest that requires an iliac crest wound catheter

Exclusion Criteria:

* Patient or parent/guardian refusal
* Ropivacaine allergy

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients that require an iliac crest bone harvest that requires an iliac crest wound catheter
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2015-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Unbound serum ropivicaine levels at postoperative day 0, 1, and 3 | three days
  Three blood draws

SECONDARY OUTCOMES:
Pain scores | Three days
  Measure of pain scores for the first three postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Franklyn Cladis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- The Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
If the participants would like to see their individual data, they may. If the data demonstrates that their plasma local anesthetic levels were high we will notify the participants and their guardians.